CLINICAL TRIAL: NCT02864030
Title: Multicenter, Interventional, Single-arm, Phase IV Study Evaluating Tolerability of Eribulin and Its Relationship With a Set of Polymorphisms in an Unselected Population of Female Patients With Metastatic Breast Cancer
Brief Title: PAINTER: Polymorphism And INcidence of Toxicity in ERibulin Treatment
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Oncologia Medica dell'Ospedale Fatebenefratelli (Other Government)
Collaborators: Mario Negri Institute for Pharmacological Research (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: PAINTER01
Record Dates: First submitted 2016-08-03; First posted 2016-08-11 (Estimated); Last update posted 2021-03-04 (Actual); Status verified 2021-03

CONDITIONS: Metastatic Breast Cancer; Toxicity; Neurotoxicity; Drug Toxicity; Adverse Drug Event
Keywords: Eribulin mesylate; Halaven; Polymorphisms; Tolerability
MeSH Terms: conditions — Breast Neoplasms; Neurotoxicity Syndromes; Drug-Related Side Effects and Adverse Reactions | interventions — eribulin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Single arm with Eribulin mesylate (Other)
  Interventions: Drug: ERIBULIN MESYLATE

INTERVENTIONS:
Drug: ERIBULIN MESYLATE — Eribulin mesylate will be administered according to the European Medicines Agency (EMA) and Italian Medicines Agency (AIFA) approved indications and schedule consists in 1.23 mg/m2 on day 1 and on day 8 of each cycle. Cycles will be repeated every 21 days until progression of disease, unacceptable toxicity, patient refusal or medical decision.
  The decision to treat patients with Eribulin is independent from the trial. Patients will be treated and managed according to clinical practice. The physician can choose any further line of treatment after disease progression with Eribulin.
  Other Names: HALAVEN

SUMMARY:
On March 17th, 2011, the European Commission issued a marketing authorization valid throughout the European Union for Eribulin mesylate (Halaven; Eisai Limited), for the treatment of patients with locally advanced or metastatic breast cancer who have progressed after at least two chemotherapic regimens for advanced disease.

As the use of Eribulin will be widespread in this tumor setting, a better knowledge of its safety profile outside clinical trials is warranted.

Indeed the possibility to select patients at risk for developing Eribulin-induced neuropathy, will allow the exclusion from these treatment of those patients harbouring the specific single nucleotide polymorphism (SNP). Given that Eribulin toxicity often results in treatment discontinuation, the ability to anticipate which patients will experience severe toxicity could allow for either early intervention or even possibly for prophylactic therapy, or for selection of the patients to be treated.

DETAILED DESCRIPTION:
This study is primarily aimed at surveying the tolerability profile of Eribulin in an unselected population of patients with metastatic breast cancer in relation to toxicities already described in clinical trials, and neurotoxicity in particular.

The secondary objectives of this trial include:

* To study the relationship between specific genetic polymorphism and incidence and severity of peripheral neuropathy
* To describe treatment efficacy in terms of duration of treatment and impact on survival.

All toxicities will be collected and classified according to National Cancer Institute Common Terminology criteria for Adverse Events (NCI CTCAE) version 4.0 and monitored during all the treatment period and up to 30 days after therapy discontinuation.

In particular, evaluation of incidence and outcome of any grade AEs already recorded in previous clinical trials will be collected, as follows:

* asthenia/fatigue,
* neutropenia,
* alopecia,
* nausea,
* peripheral neuropathy
* constipation

Any other unexpected AEs shall be evaluated likewise.

Patients must be followed for AEs until every ongoing Eribulin-related/unrelated toxicity and AE have been resolved, or the Investigator assesses them as "chronic" or "stable" or until the end of the trial, whichever comes first. For patients who will begin a new anticancer therapy after the last study drug administration, the AEs reporting period will end at the time the new treatment starts.

For the determination of polymorphisms, a routine blood collection of two tubes with 3-5 ml of blood be performed. The sample can be collected at any time during the participant's first two treatment cycles. Blood will be collected in a Vacutainer containing ethylendiaminetetraacetic acid (EDTA). Immediately after blood collection, tubes have to be inverted (at least five times) and then stored at - 20° C.

ELIGIBILITY:
Inclusion Criteria:

* Diagnosis of metastatic breast cancer
* Previous treatment with anthracyclines and taxanes
* Patients who will start Eribulin or who have already received only the first dose (cycle 1, day 1) of Eribulin according to the approved indication
* Ability to comply with sample collection
* Patient has signed the study Informed Consent Form (ICF) and the specific Pharmacogenetic ICF.
* Absence of any contraindication to treatment

Exclusion Criteria:

* Previous treatment with Eribulin in a previous line of treatment
* Previous treatment with Eribulin off label

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2014-05; Primary Completion 2018-12-31 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Incidence, time of onset, severity and duration of all Adverse Events (AEs) experienced during treatment with Eribulin (any grade) | Trough study completion, an average of 1 year
  All toxicities and their grade will be reported according to Common Terminology criteria for Adverse Events (CTCAE) v4.0, especially the most common AEs reported in previous clinical studies (asthenia/fatigue, neutropenia, alopecia, nausea, peripheral neuropathy and constipation) but also other possible unexpected toxicities.
Association between a set of selected polymorphisms and the onset of any grade peripheral neuropathy | Trough study completion, an average of 1 year
  The association between a set of selected polymorphisms and the onset of all grades peripheral neuropathy will be investigated using blood samples collected at the time of treatment initiation.
Treatment tolerability | Trough study completion, an average of 1 year
  Treatment tolerability will also be described in terms of dose intensity and dose schedule maintenance.
DOT (Duration Of Treatment) | Trough study completion, an average of 1 year
  DOT will be calculated for each patient from the date of start of Eribulin treatment to the date of last Eribulin administration for any cause (i.e. progression of disease, unacceptable toxicity, patient refusal or physician decision).
OS (Overall Survival) | Trough study completion, an average of 1 year
  OS will be calculated from the date of start of therapy to the date of death.

OTHER OUTCOMES:
The European Organization for research and treatment of cancer Quality of Life Questionnaire EORTC QLQ - C30 | Trough study completion, an average of 1 year
  This is a kind of assessment to evaluate the quality of life of cancer patients during Eribulin treatment using unique measurements that share a common Unit of Measure
Breast Cancer-Specific Quality of Life Questionnaire QlQ - BR23 | Trough study completion, an average of 1 year
  This is a kind of assessment to evaluate the quality of life during Eribulin treatment using unique measurements that share a common Unit of Measure

CONTACTS AND LOCATIONS:
Overall Officials: Laboratory of Clinical Research Department of Oncology IRCCS, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri; Giovanna Damia, PHD, Study Chair — Istituto Di Ricerche Farmacologiche Mario Negri
Locations (20):
- Italy (20):
  - Comprensorio sanitario di Bolzano, Bolzano
  - Istituti Ospitalieri di Cremona, Cremona
  - Azienda Ospedaliera S. Croce e Carle, Cuneo
  - A.O.U. Careggi, Florence
  - A.O. Vito Fazzi, Lecce
  - Ospedale Civile di Legnano, Legnano
  - Oncologia Medica Ospedale Fatebenefratelli, Milan
  - ASL Salerno Presidio Ospedaliero Andrea Tortora, Pagani
  - Fondazione IRCCS Policlinico San Matteo di Pavia, Pavia
  - Azienda Ospedaliera di Piacenza, Piacenza
  - POliclinico Universitario Campus Bio-Medico, Roma
  - Fondazione Policlinico Tor Vergata, Roma
  - Istituto Nazionale Tumori "Regina Elena" Oncologia Medica A, Roma
  - Istituto Nazionale Tumori "Regina Elena" Oncologia medica B, Roma
  - Policlinico Universitario Agostino Gemelli, Roma
  - Azienda Ospedaliera Valtellina e Valchiavenna - Presidio di Sondrio, Sondrio
  - ASL di FRosinone Ospedale SS Trinità di Sora, Sora
  - A.O. Santa Maria di Terni, Terni
  - Ospedale di Treviglio, Treviglio
  - Azienda Ospedaliero-Universitaria Santa Maria della Misericordia, Udine

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Guarneri V, Conte PF. The curability of breast cancer and the treatment of advanced disease. Eur J Nucl Med Mol Imaging. 2004 Jun;31 Suppl 1:S149-61. doi: 10.1007/s00259-004-1538-5. Epub 2004 Apr 24. PMID 15107948
- [Background] Mauri D, Polyzos NP, Salanti G, Pavlidis N, Ioannidis JP. Multiple-treatments meta-analysis of chemotherapy and targeted therapies in advanced breast cancer. J Natl Cancer Inst. 2008 Dec 17;100(24):1780-91. doi: 10.1093/jnci/djn414. Epub 2008 Dec 9. PMID 19066278
- [Background] Kobayashi T, Ichiba T, Sakuyama T, Arakawa Y, Nagasaki E, Aiba K, Nogi H, Kawase K, Takeyama H, Toriumi Y, Uchida K, Kobayashi M, Kanehira C, Suzuki M, Ando N, Natori K, Kuraishi Y. Possible clinical cure of metastatic breast cancer: lessons from our 30-year experience with oligometastatic breast cancer patients and literature review. Breast Cancer. 2012 Jul;19(3):218-37. doi: 10.1007/s12282-012-0347-0. Epub 2012 Apr 25. PMID 22532161
- [Background] Jordan MA, Kamath K, Manna T, Okouneva T, Miller HP, Davis C, Littlefield BA, Wilson L. The primary antimitotic mechanism of action of the synthetic halichondrin E7389 is suppression of microtubule growth. Mol Cancer Ther. 2005 Jul;4(7):1086-95. doi: 10.1158/1535-7163.MCT-04-0345. PMID 16020666
- [Background] Okouneva T, Azarenko O, Wilson L, Littlefield BA, Jordan MA. Inhibition of centromere dynamics by eribulin (E7389) during mitotic metaphase. Mol Cancer Ther. 2008 Jul;7(7):2003-11. doi: 10.1158/1535-7163.MCT-08-0095. PMID 18645010
- [Background] Towle MJ, Salvato KA, Budrow J, Wels BF, Kuznetsov G, Aalfs KK, Welsh S, Zheng W, Seletsky BM, Palme MH, Habgood GJ, Singer LA, Dipietro LV, Wang Y, Chen JJ, Quincy DA, Davis A, Yoshimatsu K, Kishi Y, Yu MJ, Littlefield BA. In vitro and in vivo anticancer activities of synthetic macrocyclic ketone analogues of halichondrin B. Cancer Res. 2001 Feb 1;61(3):1013-21. PMID 11221827
- [Background] Goel S, Mita AC, Mita M, Rowinsky EK, Chu QS, Wong N, Desjardins C, Fang F, Jansen M, Shuster DE, Mani S, Takimoto CH. A phase I study of eribulin mesylate (E7389), a mechanistically novel inhibitor of microtubule dynamics, in patients with advanced solid malignancies. Clin Cancer Res. 2009 Jun 15;15(12):4207-12. doi: 10.1158/1078-0432.CCR-08-2429. Epub 2009 Jun 9. PMID 19509177
- [Background] Tan AR, Rubin EH, Walton DC, Shuster DE, Wong YN, Fang F, Ashworth S, Rosen LS. Phase I study of eribulin mesylate administered once every 21 days in patients with advanced solid tumors. Clin Cancer Res. 2009 Jun 15;15(12):4213-9. doi: 10.1158/1078-0432.CCR-09-0360. Epub 2009 Jun 9. PMID 19509146
- [Background] Mukohara T, Nagai S, Mukai H, Namiki M, Minami H. Eribulin mesylate in patients with refractory cancers: a Phase I study. Invest New Drugs. 2012 Oct;30(5):1926-33. doi: 10.1007/s10637-011-9741-2. Epub 2011 Sep 2. PMID 21887501
- [Background] Vahdat LT, Pruitt B, Fabian CJ, Rivera RR, Smith DA, Tan-Chiu E, Wright J, Tan AR, Dacosta NA, Chuang E, Smith J, O'Shaughnessy J, Shuster DE, Meneses NL, Chandrawansa K, Fang F, Cole PE, Ashworth S, Blum JL. Phase II study of eribulin mesylate, a halichondrin B analog, in patients with metastatic breast cancer previously treated with an anthracycline and a taxane. J Clin Oncol. 2009 Jun 20;27(18):2954-61. doi: 10.1200/JCO.2008.17.7618. Epub 2009 Apr 6. PMID 19349550
- [Background] Cortes J, Vahdat L, Blum JL, Twelves C, Campone M, Roche H, Bachelot T, Awada A, Paridaens R, Goncalves A, Shuster DE, Wanders J, Fang F, Gurnani R, Richmond E, Cole PE, Ashworth S, Allison MA. Phase II study of the halichondrin B analog eribulin mesylate in patients with locally advanced or metastatic breast cancer previously treated with an anthracycline, a taxane, and capecitabine. J Clin Oncol. 2010 Sep 1;28(25):3922-8. doi: 10.1200/JCO.2009.25.8467. Epub 2010 Aug 2. PMID 20679609
- [Background] Aogi K, Iwata H, Masuda N, Mukai H, Yoshida M, Rai Y, Taguchi K, Sasaki Y, Takashima S. A phase II study of eribulin in Japanese patients with heavily pretreated metastatic breast cancer. Ann Oncol. 2012 Jun;23(6):1441-8. doi: 10.1093/annonc/mdr444. Epub 2011 Oct 11. PMID 21989327
- [Background] Cortes J, O'Shaughnessy J, Loesch D, Blum JL, Vahdat LT, Petrakova K, Chollet P, Manikas A, Dieras V, Delozier T, Vladimirov V, Cardoso F, Koh H, Bougnoux P, Dutcus CE, Seegobin S, Mir D, Meneses N, Wanders J, Twelves C; EMBRACE (Eisai Metastatic Breast Cancer Study Assessing Physician's Choice Versus E7389) investigators. Eribulin monotherapy versus treatment of physician's choice in patients with metastatic breast cancer (EMBRACE): a phase 3 open-label randomised study. Lancet. 2011 Mar 12;377(9769):914-23. doi: 10.1016/S0140-6736(11)60070-6. Epub 2011 Mar 2. PMID 21376385
- [Background] Cavaletti G, Alberti P, Marmiroli P. Chemotherapy-induced peripheral neurotoxicity in the era of pharmacogenomics. Lancet Oncol. 2011 Nov;12(12):1151-61. doi: 10.1016/S1470-2045(11)70131-0. Epub 2011 Jun 28. PMID 21719347
- [Background] Swain SM, Arezzo JC. Neuropathy associated with microtubule inhibitors: diagnosis, incidence, and management. Clin Adv Hematol Oncol. 2008 Jun;6(6):455-67. PMID 18567992
- [Background] Baldwin RM, Owzar K, Zembutsu H, Chhibber A, Kubo M, Jiang C, Watson D, Eclov RJ, Mefford J, McLeod HL, Friedman PN, Hudis CA, Winer EP, Jorgenson EM, Witte JS, Shulman LN, Nakamura Y, Ratain MJ, Kroetz DL. A genome-wide association study identifies novel loci for paclitaxel-induced sensory peripheral neuropathy in CALGB 40101. Clin Cancer Res. 2012 Sep 15;18(18):5099-109. doi: 10.1158/1078-0432.CCR-12-1590. Epub 2012 Jul 27. PMID 22843789
- [Background] Sucheston LE, Zhao H, Yao S, Zirpoli G, Liu S, Barlow WE, Moore HC, Thomas Budd G, Hershman DL, Davis W, Ciupak GL, Stewart JA, Isaacs C, Hobday TJ, Salim M, Hortobagyi GN, Gralow JR, Livingston RB, Albain KS, Hayes DF, Ambrosone CB. Genetic predictors of taxane-induced neurotoxicity in a SWOG phase III intergroup adjuvant breast cancer treatment trial (S0221). Breast Cancer Res Treat. 2011 Dec;130(3):993-1002. doi: 10.1007/s10549-011-1671-3. Epub 2011 Jul 16. PMID 21766209
- [Background] Mir O, Alexandre J, Tran A, Durand JP, Pons G, Treluyer JM, Goldwasser F. Relationship between GSTP1 Ile(105)Val polymorphism and docetaxel-induced peripheral neuropathy: clinical evidence of a role of oxidative stress in taxane toxicity. Ann Oncol. 2009 Apr;20(4):736-40. doi: 10.1093/annonc/mdn698. Epub 2009 Feb 17. PMID 19223573
- [Background] Sissung TM, Mross K, Steinberg SM, Behringer D, Figg WD, Sparreboom A, Mielke S. Association of ABCB1 genotypes with paclitaxel-mediated peripheral neuropathy and neutropenia. Eur J Cancer. 2006 Nov;42(17):2893-6. doi: 10.1016/j.ejca.2006.06.017. Epub 2006 Sep 6. PMID 16950614
- [Background] Hasmats J, Kupershmidt I, Rodriguez-Antona C, Su QJ, Khan MS, Jara C, Mielgo X, Lundeberg J, Green H. Identification of candidate SNPs for drug induced toxicity from differentially expressed genes in associated tissues. Gene. 2012 Sep 10;506(1):62-8. doi: 10.1016/j.gene.2012.06.053. Epub 2012 Jul 1. PMID 22759513
- [Background] Johnson DC, Corthals SL, Walker BA, Ross FM, Gregory WM, Dickens NJ, Lokhorst HM, Goldschmidt H, Davies FE, Durie BG, Van Ness B, Child JA, Sonneveld P, Morgan GJ. Genetic factors underlying the risk of thalidomide-related neuropathy in patients with multiple myeloma. J Clin Oncol. 2011 Mar 1;29(7):797-804. doi: 10.1200/JCO.2010.28.0792. Epub 2011 Jan 18. PMID 21245421
- [Derived] La Verde N, Damia G, Garrone O, Santini D, Fabi A, Ciccarese M, Generali DG, Nunzi M, Poletto E, Ferraris E, Cretella E, Scandurra G, Meattini I, Bertolini AS, Cavanna L, Collova E, Romagnoli E, Rulli E, Legramandi L, Guffanti F, Bramati A, Moretti A, Cassano A, Vici P, Torri V, Farina G; PAINTER investigators. Tolerability of Eribulin and correlation between polymorphisms and neuropathy in an unselected population of female patients with metastatic breast cancer: results of the multicenter, single arm, phase IV PAINTER study. Breast Cancer Res. 2022 Oct 28;24(1):71. doi: 10.1186/s13058-022-01560-w. PMID 36307826